CLINICAL TRIAL: NCT05950763
Title: The Causes of Academic Excellence Concentrated in Dormitory
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Zhejiang Chinese Medical University (Other Government)
Responsible Party: Principal Investigator, Ying Xu, prime investigator, Zhejiang Chinese Medical University
Other Study IDs: 20230427-2
Record Dates: First submitted 2023-06-06; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Peer Influence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research will take the sophomore to senior students of Zhejiang University of Traditional Chinese Medicine as the research object to investigate the influence of dormitory atmosphere on the academic performance, scientific research achievements, and competition awards of dormitory members, analyze the path of straightforward-A student dormitory formation, and find out the current Weak links of college students' ideological and political education in dormitory culture construction, and explore how dormitory culture construction can promote the common progress of dormitory members

ELIGIBILITY:
Inclusion Criteria:

* Sophomore-senior students of Zhejiang University of Traditional Chinese Medicine

Exclusion Criteria:

* Non-straight-A student dormitory member

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: It refers to two or more members in a dormitory who have achieved outstanding academic performance, have better scientific research results, have better competition awards (meet one or more), and usually study hard and study hard
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Academic Excellence Concentrated in Dormitory | Zhejiang University of Traditional Chinese Medicine sophomore-senior students from admission to September 2023
  Academic performance (required course grade points)in units of credits, scientific research achievements are indexed by the number of papers produced, competition awards are based on the number of awards won,dormitory atmosphere is based on the combined score of each option of the questionnaire as an indicator（A is 0 points, B is 5 points……）

CONTACTS AND LOCATIONS:
Locations (1):
- Ying Xu, Hangzhou, Zhejiang, China